CLINICAL TRIAL: NCT02250885
Title: Investigator Initiated, Phase 2 Clinical Trial of Selinexor (KPT-330) for the Treatment of Poorly Differentiated Lung and Gastroenteropancreatic Tumors
Brief Title: KPT-330 to Treat Poorly Differentiated Lung and Gastroenteropancreatic Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gabrail Cancer Center Research (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCC-003
Record Dates: First submitted 2014-08-21; First posted 2014-09-26 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Carcinoma, Neuroendocrine
Keywords: Selinexor; phase 2; Gabrail
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selinexor (KPT-330) (Experimental): Selinexor will be taken orally at a starting dose of 50mg/m2 twice weekly on weeks 1, 2, and 3 of each 4 week cycle.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Selective Inhibitor fo Nuclear Export (SINE)
  Other Names: KPT-330

SUMMARY:
Evaluate the efficacy of Selinexor in patients with poorly differentiated lung and gastrointestinal and pancreatic neuroendocrine tumors.

DETAILED DESCRIPTION:
Evaluate the efficacy of Selinexor in patients with poorly differentiated lung and gastrointestinal and pancreatic neuroendocrine tumors in adult patients age >/= to 18.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with federal, local, and institutional guidelines
* Age ≥18 years
* Patients must have a tissue diagnosis of any of the following:

  * Small cell lung cancer (SCLC) or poorly differentiated gastroenteropancreatic neuroendocrine tumor (GEP-NET)
  * Poorly differentiated metastatic neuroendocrine tumors of unknown primary origin
* Measurable disease: Any primary and/or metastatic mass reproducibly measurable in one or two diameters by RECIST 1.1 parameters by cat scan (CT) scan.
* Objective evidence of tumor progression within 4 months prior to study entry, as defined by serial cat scan (CT) per RECIST 1.1 criteria. (At least a 20% increase in the sum of diameters of target lesions. In addition, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression).
* Patients must have received at least one prior line of chemotherapy and must have exhausted any other standard-of-care treatment option.
* Prior radiation and surgery is allowed. At least 3 weeks should have elapsed from surgery, chemotherapy, hepatic embolization/ chemoembolization or radioactive isotopes (i.e. Yttrium 90). In any case, disease progression must be documented after treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Concomitant octreotide treatment for carcinoid syndrome is allowed for patients whose tumor has progressed while on octreotide. Patients must have been on a stable dose of octreotide two weeks prior to enrollment and must remain on a stable dose during the study.
* Hematological function:

  * Total white blood cell count (WBC) > 2,000/mm³
  * Absolute neutrophil (ANC) > 1,000/mm³
  * Platelet >100,000mm³
* Adequate hepatic function within 14 days prior to C1D1: total direct bilirubin <2 times the upper limit of normal (ULN; 1.0 mg/dL) and alanine aminotransferase (ALT) <2.5 times ULN (30 U/L). In the case of known (radiological and/or biopsy documented) liver metastasis, ALT <5.0 times ULN is acceptable.
* Adequate renal function within 7 days prior to C1D1: estimated creatinine clearance of ≥ 30 mL/min, calculated using the formula of Cockcroft and Gault: (140-Age) • Mass (kg)/(72 • creatinine mg/dL); multiply by 0.85 if female.
* Blood electrolytes should be within the following normal limits:

Bicarbonate (total) 18-30 mEq/L Sodium 135-147 mEq/L Potassium 3.5-5.5 mEq/L Phosphorus 1.8-2.3 mEq/L Magnesium 1.5-3.0 mEq/L Chloride 98-106 mEq/L Calcium (total) 4.5-5.5 mEq/L

* Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose.

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients with the following tumor types: lung carcinoid, pheochromocytomas, paragangliomas, medullary thyroid carcinomas, any other tumors with neuroendocrine features not listed in the inclusion criteria
* Radiation, chemotherapy, or immunotherapy or any other anticancer therapy ≤3 weeks prior to C1D1
* Major surgery ≤3 weeks prior to C1D1
* Unstable cardiovascular function:

  * Congestive heart failure (CHF) of NYHA Class ≥3 OR
  * Myocardial infarction (MI) within 3 months
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; patients with controlled infection or on prophylactic antibiotics are permitted in the study
* Known to be human immunodeficiency virus (HIV) seropositive
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV RNA) or HBsAg (HBV surface antigen)
* Any underlying condition that would significantly interfere with the absorption of an oral medication
* Patients who have active central nervous system (CNS) malignancy. Asymptomatic small lesions are not considered active. Treated lesions may be considered inactive if they are stable for at least 3 months. Patient with malignant cells in their cerebrospinal fluid (CSF) without CNS symptom may be included.
* Serious psychiatric or medical conditions that could interfere with treatment
* Patients with coagulation problems and active bleeding in the last month (peptic ulcer, epistaxis, spontaneous bleeding)
* Patients with signs of gastrointestinal obstruction or uncontrolled vomiting or diarrhea (>3 episodes/week) with electrolyte abnormalities
* Concurrent therapy with approved or investigational anticancer therapeutic agents other than glucocorticoids
* Participation in an investigational anti-cancer study within 3 weeks prior to cycle 1 day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Every 8 weeks from screening until documented disease progression or date of death, whichever occurs first, up to approximately 100 months.
  To evaluate the efficacy of single agent Selinexor in patients with poorly differentiated lung and gastroenteropancreatic (GEP) neuroendocrine tumors (NET) as determined by overall response rate (ORR) including complete (CR) and partial (PR) response.

CONTACTS AND LOCATIONS:
Overall Officials: Nashat Y Gabrail, MD, Principal Investigator — Gabrail Cancer Center Research
Locations (1):
- Gabrail Cancer Center Research, Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No